CLINICAL TRIAL: NCT01273272
Title: Cognitive-Behavioral Treatment for Patients With Mild Alzheimer's Dementia: A Randomized Controlled Trial
Brief Title: Cognitive-Behavioral Treatment for Mild Alzheimer's Patients and Their Caregivers
Acronym: CBTAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Simon Forstmeier, Ph.D., University of Zurich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-130034/1a
Record Dates: First submitted 2011-01-03; First posted 2011-01-10 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Alzheimer Disease
Keywords: Cognitive Behavior Therapy; Early dementia, Alzheimer type
MeSH Terms: conditions — Alzheimer Disease | interventions — Psychosocial Intervention; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (CBT) (Experimental): Comprehensive, CBT-based, multi-component treatment. Comprehensive CBT intervention in addition to standard treatment
  Interventions: Behavioral: Comprehensive, CBT-based, multi-component treatment
- Treatment as usual (TAU) (Active Comparator): Standard Treatment (medical and psychosocial)
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Comprehensive, CBT-based, multi-component treatment — It includes eight modules: diagnosis and goal setting; psychoeducation; engagement in pleasant activities; cognitive restructuring; live review; training caregiver in behavior man-agement techniques; interventions for the caregiver; and couples counselling. It consists of 20 weekly sessions (plus appr. 5 single session with caregiver).
  Other Names: Psychosocial intervention
  Arms: Cognitive Behavioral Therapy (CBT)
Behavioral: Treatment as usual — Each patient/caregiver must receive at least three out of six interventions: (1) psychoeducation on dementia and treatment of dementia (oral and written); (2) appropriate medical treatment; (3) social counseling by specialized staff; (4) memory training in group setting; (5) self-help group for the patient; (6) self-help group for the caregiver.
  Other Names: Standard treatment
  Arms: Treatment as usual (TAU)

SUMMARY:
The purpose of this study is to determine whether a comprehensive cognitive-behavioral therapy-based, multi-component treatment programme is effective in the treatment of neuropsychiatric symptoms of patients with mild Alzheimer's dementia.

DETAILED DESCRIPTION:
Mild Alzheimer's dementia (AD) cases are with 15 millions worldwide the largest fraction of all AD cases. Most patients are cared for by their family at home. Neuropsychiatric symptoms are very common in AD, even as early as in mild AD: About 90% of all mild AD cases experience neuropsychiatric symptoms, most frequently depression, anxiety, and irritability. These symptoms are associated with greater morbidity, reduced quality of life for the patient, increased burden and depression for the caregiver, higher costs of care, and nursing home placement. Thus, interventions aimed at treating these symptoms could have a tremendous effect on pa-tients, caregivers, and society.

This study is a randomized, controlled trial (RCT) evaluating a comprehensive CBT-based, multi-component treatment programme consisting of eight modules (diagnosis and goal-setting; psycho-education; engagement in pleasant activities; cognitive restructuring; life review; training caregiver in behavior management techniques; interventions for the caregiver; couples counseling) and 20 sessions.

This trial aims at significantly reducing depressive and other neuropsychiatric symptoms in the AD patients, and secondary in reducing burden and depressive symptoms of the caregivers. Patients with AD alone or mixed AD and vascular dementia that are in the mild stage and suffer under any neuropsychiatric symptom will be included. The patients and their caregiver will be randomized to either the CBT-based intervention or to the control condition that receives treatment as usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

* Patients have to meet NINCDS-ADRDA criteria for probable or possible AD (McKhann et al., 1984). Mixed Alzheimer and Vascular dementia cases will also be included.
* Only AD cases with a mild dementia severity will be included, determined by the Clinical Dementia Rating (CDR) scale (i.e. scores of 0.5 or 1, Morris, 1993) and by the Mini Mental State Examination (MMSE) (i.e. scores of 20 or more, Folstein, Folstein, & McHugh, 1975).
* The patient must suffer under any non-cognitive symptom that motivates him to accept psy-chotherapeutic help.
* A caregiver must be available to take part in most of the therapy sessions.

Exclusion Criteria:

* concomitant alcohol or drug addiction and a history of a malignant disease, severe organ failure, metabolic or hematologic disorders, neurosurgery or neurological condition such as Parkinson's disease, epilepsy, postencephalitic and postconcussional syndrome

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Geriatric Depression Scale (GDS) | Pre-treatment, posttreatment (expected average of 9 months after protreatment), 6- and 12-months follow-up

SECONDARY OUTCOMES:
Change from baseline in Neuropsychiatric Inventory (NPI) | Pre-treatment, post-treatment (expected average of 9 months after protreatment), 6- and 12-months follow-up
Change from baseline in Bayer-Activities of Daily Living (B-ADL) | Pre-treatment, post-treatment (expected average of 9 months after protreatment), 6- and 12-months follow-up
Change from baseline in Stress Coping Inventory (SCI) | Pre-treatment, post-treatment (expected average of 9 months after protreatment), 6- and 12-months follow-up
Change from baseline in Apathy Evaluation Scale (AES) | Pre-treatment, post-treatment (expected average of 9 months after protreatment), 6- and 12-months follow-up
Caregiver: Change from baseline in Center for Epidemiologic Studies Depression Scale (CES-D) | Pre-treatment, post-treatment (expected average of 9 months after protreatment), 6- and 12-months follow-up
Caregiver: Change from baseline in Trait scale of the State Trait Anxiety Inventory (STAI) | Pre-treatment, post-treatment (expected average of 9 months after protreatment), 6- and 12-months follow-up
Caregiver: Change from baseline in Anger-in and anger-out scales of the State Trait Anger Expression Inventory (STAXI) | Pre-treatment, post-treatment (expected average of 9 months after protreatment), 6- and 12-months follow-up
Caregiver: Change from baseline in Short-Form Health Survey (SF-12) | Pre-treatment, post-treatment (expected average of 9 months after protreatment), 6- and 12-months follow-up
Caregiver: Change from baseline in Zarit Burden Interview (ZBI) | Pre-treatment, post-treatment (expected average of 9 months after protreatment), 6- and 12-months follow-up
Caregiver: Change from baseline in Stress Coping Inventory (SCI) | Pre-treatment, post-treatment (expected average of 9 months after protreatment), 6- and 12-months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Simon Forstmeier, Ph.D., Principal Investigator — University of Zurich; Andreas Maercker, M.D.,Ph.D., Study Chair — University of Zurich; Egemen Savaskan, M.D., Study Chair — Psychiatric University Hospital, Zurich; Tanja Roth, Ph.D., Study Chair — Psychiatric University Hospital, Zurich
Locations (1):
- Psychiatric University Hospital, Clinic for Geriatric Medicine, Zurich, Switzerland

REFERENCES:
- [Background] Forstmeier S, Maercker A. Problems of aging. Psychotherapy in older age [German]. Göttingen, Germany: Hogrefe. 2008.
- [Background] Forstmeier S, Maercker A. Psychotherapie im Alter. Psychotherapeutenjournal 4: 340-352, 2007
- [Background] Forstmeier S, Maercker A, Savaskan E, Roth T. Cognitive behavioural treatment for mild Alzheimer's patients and their caregivers (CBTAC): study protocol for a randomized controlled trial. Trials. 2015 Nov 17;16:526. doi: 10.1186/s13063-015-1043-0. PMID 26576633
- [Derived] Forstmeier S, Maercker A, Bohli L, Savaskan E, Roth T. Cognitive behavioural treatment for mild Alzheimer's patients and their caregivers (CBTAC): results of a randomised controlled trial. Aging Ment Health. 2025 Feb;29(2):359-368. doi: 10.1080/13607863.2024.2393748. Epub 2024 Aug 20. PMID 39164933